CLINICAL TRIAL: NCT03972111
Title: A Phase 4, Observational Field Study to Evaluate the Safety and Clinical Benefit of TPOXX (Tecovirimat)-Treated Patients Following Exposure to Variola Virus and Clinical Diagnosis of Smallpox Disease
Brief Title: A Phase 4, Observational Field Study to Evaluate TPOXX in Patients With Smallpox
Status: Withdrawn | Type: Observational
Why Stopped: commitment fulfilled
Sponsor: SIGA Technologies (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: SIGA-246-021
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Smallpox
MeSH Terms: conditions — Smallpox | interventions — tecovirimat

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — smallpox lesion samples and blood collected to assess viral DNA levels and conduct genotypic resistance analysis and phenotypic analysis if possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: TPOXX 200Mg Capsule — TPOXX 600 mg (three 200 mg.) capsules twice daily for 14 days
  Other Names: tecovirimat

SUMMARY:
Phase 4, Observational Field Study in Patients Treated With TPOXX for Smallpox Disease

DETAILED DESCRIPTION:
Phase 4, Observational Field Study to evaluate safety and clinical benefit of TPOXX (tecovirimat) in patients treated with TPOXX following exposure to variola virus and a clinical diagnosis of smallpox disease.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent or assent themselves or through a guardian or legally authorized representative, receiving or initiating treatment with TPOXX, and willing and able to adhere to the recommended procedures in the protocol.
* Determined, per the clinical definition of smallpox, that the patient presenting with a case of acute, generalized vesicular/pustular rash meets Centers for Disease Control and Prevention (CDC) criteria of having confirmed, suspected, or probable smallpox and/or is at high or moderate risk for developing smallpox.
* The CDC in coordination with the Department of Health and Human Services/Assistant Secretary for Preparedness and Response (ASPR) has released TPOXX to the physician or designated health authorities for patient treatment, and the CDC has provided physician contact information to PPD, the contract research organization.

Exclusion Criteria:

• Known allergy to tecovirimat and/or excipients of TPOXX.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric patients who weigh ≥13 kg who receive FDA-approved TPOXX as part of their medical treatment for variola virus (VARV) infection in the United States (US). These patients will have suspected, probable, or confirmed smallpox. The purpose of this field study is to evaluate the safety, survival status, time to death, and smallpox rash progression in patients who are receiving TPOXX for the treatment of smallpox in the US
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Assess survival | 44 days post first dose of TPOXX
  To assess the overall survival at Day 44 following treatment with TPOXX

SECONDARY OUTCOMES:
Survival status | 14 days post first dose of TPOXX
  Survival status after completion of 14 days of TPOXX treatment will be assessed by physician for inpatients and collected from patient via patient diary question or follow up telephone contact.
Time to death | From date of treatment with TPOXX until the date of death from any cause, whichever came first, assessed up to 44 days after TPOXX treatment
  Time to death after treatment with TPOXX

OTHER OUTCOMES:
Exploratory objective-TPOXX plasma concentration | Plasma samples will be collected to determine the plasma concentration of TPOXX from Days 1-14 of the TPOXX treatment period for inpatients. This data will be reported.
  To evaluate the plasma concentration of TPOXX from any available samples

CONTACTS AND LOCATIONS:
Overall Officials: Dennis E. Hruby, PhD, Study Director — SIGA Technologies
Locations (1):
- Investigator Site, Corvallis, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided